CLINICAL TRIAL: NCT00832663
Title: The Influence of Blocking Inflammatory Activity in Vivo on Skeletal Muscle Regeneration in Humans
Brief Title: Influence of Non-steroidal Anti-inflammatory Drugs (NSAID) on Muscle Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Lundbeck Foundation (Other); Team Denmark (Other); Danish Ministry of Culture (Unknown); Anti Doping Danmark (Other); The Danish Rheumatism Association (Other); King Christian IX and Queen Louise Jubilee Bursary (Unknown)
Responsible Party: Abigail Mackey, Institute of Sports Medicine Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AM_P64_BBH; H-D-2008-074
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Muscle Damage
Keywords: Muscle regeneration; Satellite cells; electrical stimulation; eccentric contractions; myogenic precursor cells
MeSH Terms: interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NSAID (Experimental): receive NSAID
  Interventions: Drug: NSAID
- Placebo (Placebo Comparator): receive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NSAID — Effect of NSAID ingestion on muscle regeneration
  Arms: NSAID
Drug: placebo — receive placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the influence of non-steroidal anti-inflammatory drugs (NSAIDs) on muscle regeneration.

The investigators' hypothesis is that ingestion of NSAID will delay or impair muscle regeneration.

DETAILED DESCRIPTION:
The model employed to induce muscle damage is electrical stimulation. Muscle biopsies will be examined to follow the response of satellite cells and muscle regeneration. Study participants will be randomly assigned to a placebo or NSAID group in a double-blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy
* does not exercise regularly

Exclusion Criteria:

* displays contraindications for taking NSAID
* well-trained

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Muscle regeneration | 1 month

SECONDARY OUTCOMES:
Muscle strength | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Abigail L Mackey, PhD, Principal Investigator — Institute of Sports Medicine Copenhagen, Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, NV, Denmark